CLINICAL TRIAL: NCT01915927
Title: A Phase 1 Study of Autologous Mesenchymal Stromal Cell Coated Fistula Plug in Patients With Fistulizing Crohn's Disease.
Brief Title: Stem Cell Fistula Plug in Perianal Crohn's Disease
Acronym: MSC-AFP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: William A. Faubion, M.D. (Other)
Responsible Party: Sponsor-Investigator, William A. Faubion, M.D., PI, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-009716
Record Dates: First submitted 2013-07-31; First posted 2013-08-05 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Perianal Crohn's Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Only 1 arm: treatment with MSC-AFP
  Interventions: Drug: MSC-AFP

INTERVENTIONS:
Drug: MSC-AFP

SUMMARY:
The investigators propose to study the safety of autologous mesenchymal stromal cell transfer using a biomatrix (the Gore® Bio-A®; Fistula Plug) in a Phase I study using a single dose of 20 million cells. Twenty adult patients (age 18 years or older) with refractory, complicated perianal fistulizing Crohn's disease will be enrolled. Subjects will undergo standard adjuvant therapy including drainage of infection and placement of a draining seton with continuation of pre-existing anti-Crohn's therapy. Six weeks post placement of the draining seton, the seton will be replaced with the MSC loaded Gore® Bio-A® fistula plug as per current clinical practice. The subjects will be subsequently followed for fistula response and closure for 24 months. This is an autologous product derived from the patient and used only for the same patient.

ELIGIBILITY:
Inclusion Criteria

* Males and females 18-65 years of age.
* Residents of the United States.
* Crohn's disease with single or multiple draining complex perianal fistulae (definition as below) for at least three months despite standard therapy (definition below).
* Concurrent therapies with corticosteroids, 5-ASA drugs, thiopurines, MTX, antibiotics, and anti-TNF therapy are permitted.
* All patients should have undergone a colonoscopy in last 12 months to rule out malignant or premalignant condition
* Have no contraindications to MR evaluations: e.g. pacemaker or magnetically active metal fragments, claustrophobia
* Ability to comply with protocol
* Competent and able to provide written informed consent
* Must have failed standard medical therapy including anti-TNF agents

Exclusion Criteria

* Inability to give informed consent.
* Clinically significant medical conditions within the six months before administration of MSCs: e.g. myocardial infarction, active angina, congestive heart failure or other conditions that would, in the opinion of the investigators, compromise the safety of the patient.
* Specific exclusions: Evidence of hepatitis B, C, or HIV
* History of cancer including melanoma (with the exception of localized skin cancers)
* Investigational drug within thirty (30) days of baseline
* A resident outside the United States
* Pregnant or breast feeding.
* History of clinically significant auto-immunity (other than Crohn's disease) or any previous example of fat-directed autoimmunity
* Previous allergic reaction to a perianal fistula plug.
* If liposuction is not technically feasible
* Allergic to local anesthetics
* Pregnant patients or trying to become pregnant.
* Non-enterocutaneous tracts (ie recto-vaginal, entero-vesicular)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
To determine the safety and toxicity of using autologous MSC coated fistula plug in patients with fistulizing Crohn's Disease. | 2-24 months
  The primary endpoint of this study is to determine the safety and feasibility of using adipose derived, autologous mesenchymal stromal cells (MSC) bound to the Gore® Bio-A® Fistula Plug for treatment of refractory CD perianal fistulae.

SECONDARY OUTCOMES:
To assess in preliminary fashion the response of fistula healing induced by the GORE plug containing MSC | 2-24 months
  To assess in preliminary fashion the response of fistula healing induced by the GORE plug containing MSC i) Clinically by drainage assessment and ii) Radiographically by MRI, the gold standard test for assessment of healing.

CONTACTS AND LOCATIONS:
Overall Officials: William Faubion, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Dietz AB, Dozois EJ, Fletcher JG, Butler GW, Radel D, Lightner AL, Dave M, Friton J, Nair A, Camilleri ET, Dudakovic A, van Wijnen AJ, Faubion WA. Autologous Mesenchymal Stem Cells, Applied in a Bioabsorbable Matrix, for Treatment of Perianal Fistulas in Patients With Crohn's Disease. Gastroenterology. 2017 Jul;153(1):59-62.e2. doi: 10.1053/j.gastro.2017.04.001. Epub 2017 Apr 9. PMID 28400193
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials